CLINICAL TRIAL: NCT03411759
Title: Exploratory Study of Cytochrome P450's Pharmacogenomics in Chronic Pain Patients
Brief Title: Cytochrome P450's Pharmacogenomics in Chronic Pain Patients
Acronym: FACIDOCRO
Status: Completed | Type: Observational
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, Andrea Fanelli, Principal Investigator, University of Bologna
Other Study IDs: FACIDOCRO
Record Dates: First submitted 2018-01-17; First posted 2018-01-26 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2018-01

CONDITIONS: Analgesia; CYP2D6 Polymorphism; Opioid Use; Chronic Pain
Keywords: CYP2D6; Chronic pain; Cytochrome P450; Opioids
MeSH Terms: conditions — Agnosia; Chronic Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — buccal swab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The use of titrated drugs is at the base of a successful antalgic treatment in order to provide both an adequate relief and a satisfactory tolerability profile. These molecules, though, have a varying degree of efficacy in different subjects due to medical and genetic reasons. The latter are mainly represented by cytochrome (CYP) P450, in particular CYP2D6's polymorphisms are responsible for the diversified metabolism of analgesics used in chronic pain treatments.

Four main types of enzymatic metabolism make up the population, each one defined by a different CYP2D6 allele: extensive metabolizers, ultra-rapid metabolizers, intermediate metabolizers and poor metabolizers.

Moreover, regarding polytherapies, the analgesics' metabolism could be influenced by coadministration of other drugs, thus determining an inhibition or induction of the metabolic enzymes - known as phenocopying - and potentially also a change in the metabolic phenotype itself. The final outcome is the inconstancy of effectiveness and of the risk of developing side effects.

The primary objective of this study is to define a genetic pattern for the gene CYP2D6 by assessing the incidence of poor or ultrarapid metabolizers in a population of chronic pain patients. This will also allow to observe phenocopying in the same population.

Hence 100 patients diagnosed with chronic pain will be enrolled. The genetic pattern of the gene CYP2D6 of such patients will be examined by taking mouth samples. At the same time parametric tests for paired data to survey the correlations between phenotypical patterns and pharmacological therapies will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic pain

Exclusion Criteria:

-

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic pain patients who are treated in a pain therapy clinic
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2018-03-23 (Actual); Study Completion 2018-03-23 (Actual)

PRIMARY OUTCOMES:
Analyzing the genetic pattern of CYP2D6's genes | 8-10 months
  Analyzing the genetic pattern of CYP2D6's genes in a population of chronic pain patients who are treated in a pain therapy clinic

SECONDARY OUTCOMES:
Evaluating the incidence of metabolic phenotype's variation | 8-10 months
  Evaluating the incidence of metabolic phenotype's variation (phenocopying) in a population of chronic pain patients who are treated in a pain therapy clinic

CONTACTS AND LOCATIONS:
Locations (1):
- Andrea Fanelli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fanelli A, Palazzo C, Balzani E, Iuvaro A, Pelotti S, Melotti RM. An Explorative Study of CYP2D6's Polymorphism in a Sample of Chronic Pain Patients. Pain Med. 2020 May 1;21(5):1010-1017. doi: 10.1093/pm/pnz265. PMID 31710684